CLINICAL TRIAL: NCT06363513
Title: The Efficacy of Aescin in Combination With Micronized Purified Flavonoid Fraction (MPFF) in the Early Control of Bleeding From Acute Internal Hemorrhoids, A Randomized Controlled Trial
Brief Title: The Efficacy of Aescin in Combination With MPFF in the Early Control of Bleeding From Acute Internal Hemorrhoids, A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Witcha Vipudhamorn, FRCS MD, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUR2567-0150
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Anorectal Disorder
Keywords: hemorrhoid; bleeding
MeSH Terms: conditions — Rectal Diseases; Hemorrhoids; Hemorrhage | interventions — Escin; horse chestnut seed; Flavonoids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPFF with aescin group (Experimental)
  Interventions: Drug: Aescin in Horse Chestnut; Drug: Flavonoid
- MPFF group (Active Comparator)
  Interventions: Drug: Flavonoid

INTERVENTIONS:
Drug: Aescin in Horse Chestnut — Can aescin reduce bleeding in early hemorrhoid
  Arms: MPFF with aescin group
Drug: Flavonoid — Can combine aescin and MPFF reduce bleeding in early hemorrhoid
  Other Names: MPFF

SUMMARY:
Hemorrhoidal disease, characterized by symptomatic enlargement and distal displacement of anal cushions, has been a subject of recognition and management for centuries. The etymology of "hemorrhoid" is traced back to the Greek words haima (blood) and rhoos (flow). Prevalent in over 20% of the population across various life stages, this anorectal condition impacts both genders. The multifaceted development of the disease incorporates theories encompassing abnormal dilation of hemorrhoidal plexuses, distension of arteriovenous anastomoses, prolapse of anal pads, and a myriad of genetic, anatomical, dietary, and lifestyle factors. Manifestations range from venous distension to bleeding and thrombosis, with classification based on location (internal/external/combined) and degree of prolapse (grade 1-4).

Upon comprehensive history-taking and examinations, including digital rectal and proctoscope assessments, a definitive diagnosis is established, leading to the treatment phase. Although outpatient procedures demonstrate efficacy, patients may persist with pain and discomfort. Medical intervention assumes significance for stages 1 and 2, incorporating approaches such as rubber-band ligation, injection sclerotherapy, and dietary modifications. Micronized Purified Flavonoid Fraction (MPFF), integral to hemorrhoid treatment, has been scrutinized for its ability to mitigate pathogenic processes culminating in acute bleeding. The stagnation of blood in vascular plexuses prompts an inflammatory response, activating white cells and increasing vessel wall permeability. MPFF's flavonoid compounds are posited to alleviate bleeding by augmenting venous tone, reducing stasis, inhibiting inflammatory mediators, and enhancing lymphatic drainage[8]. Multiple trials substantiate MPFF's efficacy in ceasing bleeding, alleviating symptoms, and preventing hemorrhoid relapse.

Aescin, a saponin mixture found in Aesculus hippocastanum (horse chestnut). The primary active component, β-aescin, contributes to the plant's medicinal attributes. Experimental investigations in animal models underscore its anti-edematous, anti-inflammatory, and venotonic properties, attributed to molecular mechanisms facilitating ion entry into channels and elevating venous tension. While the therapeutic benefits of aescin for hemorrhoids are acknowledged, the absence of randomized control trials impedes the conclusive validation of its efficacy. In the realm of diverse treatment options, this proposed randomized controlled trial aims to assess the comparative effectiveness of combining aescin with MPFF versus MPFF alone in managing hemorrhoid-related symptoms. The study aspires to furnish valuable insights for refining therapeutic strategies in the management of hemorrhoids and enhancing patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* New case acute hemorrhoid grade 1 and 2
* Age over 18 years
* In patients aged over 50 years, it is imperative to confirm the absence of any alternative causes of bleeding through a colonoscopy
* Can long term follow up

Exclusion Criteria:

* History of bleeding disorder
* History of colorectal cancer, inflammatory bowel disease, chronic kidney disease
* Physical exam reveals anal fissure
* Pregnancy
* Any psychotic disorder
* Refuse to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Cessation of bleeding | 7 days
  day that patient no bleed of hemorrhoid

CONTACTS AND LOCATIONS:
Locations (1):
- Maharaj Chiang Mai hospital, Chiang Mai, Maung, Thailand

IPD SHARING:
Plan to Share IPD: No
published